CLINICAL TRIAL: NCT01055860
Title: One Year Outcome After Robotic Assisted Laparoscopic Sacral Colpopexy, a Case Series Review
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Patrick Culligan, MD, Atlantic Health System
Other Study IDs: R09-02-007
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence
Keywords: uterine Prolapse; vaginal prolapse; mesh erosion; urinary incontinence; bowel symptoms
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence; Uterine Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Robotic sacral colpopexy: Our study population will be women who underwent Robotic assisted laparoscopic sacral colpopexy at the Morristown Memorial Hospital for correction of pelvic organ prolapse using a synthetic polypropylene mesh.

SUMMARY:
Robotic approach to sacral colpopexy is a relatively new procedure. The literature is scarce in regard to its long-term outcomes. This advanced procedure is offered at MMH through the Urogynecology division. The Investigators setup to review the one year outcome of patients who underwent this procedure using a polypropylene mesh. These outcomes will include anatomical and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

* Any Robotic assisted laparoscopic sacral colpopexy with polypropylene mesh during the study period

Exclusion Criteria:

* Other graft material than polypropylene.
* Enrollment in a different study.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population will be women who underwent Robotic assisted laparoscopic sacral colpopexy at the Morristown Memorial Hospital for correction of pelvic organ prolapse using a synthetic polypropylene mesh.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
1. Objective anatomic outcomes We will use the pelvic organ prolapse quantification system (POP-Q). Objective surgical failure will be defined as any prolapse at or beyond the introitus | one year

SECONDARY OUTCOMES:
2. Prolapse Specific Quality of Life Patients will complete a prolapse specific quality of life instrument prior to and one year after surgery. (PFIQ-7) | one year
3. Pelvic organ prolapse related symptoms (PFDI-20) | one year
4. Graft-related complications Rates of graft erosion into adjacent organs such as bowel, bladder or vagina - during the study period will be reported. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Culligan, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Health Urogynecology, Morristown, New Jersey, United States